CLINICAL TRIAL: NCT00248144
Title: A Randomized, Multicenter, Double-Blinded Controlled Study to Compare the Effectiveness of a Single Dose (1500 mg) of Famciclovir, One Day (750 mg q12) of Famciclovir and Placebo in Patient-Initiated Episodic Treatment of Recurrent Herpes Labialis
Brief Title: A Study to Evaluate the Safety and Efficacy of Single Day or Single Dose Famciclovir for the Treatment of Recurrent Herpes Labialis
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CFAM810A2403
Record Dates: First submitted 2005-11-02; First posted 2005-11-03 (Estimated); Last update posted 2007-12-10 (Estimated); Status verified 2006-08

CONDITIONS: Recurrent Herpes Labialis
Keywords: Herpes labialis
MeSH Terms: conditions — Herpes Labialis | interventions — Famciclovir

INTERVENTIONS:
Drug: Famciclovir

SUMMARY:
The study is designed to assess the efficacy and safety of patient-initiated therapy with famciclovir 1500 mg o.d. or 750 mg b.i.d. for one day treatment in adult men and women with recurrent herpes labialis

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 18 years or older
* A history typical for recurrent herpes labialis. The subject must have experienced three or more episodes of cold sores in the last 12 months, and have a history of prodromal symptoms, as defined by the patient, preceding at least 50% of these cold sores, and must also have a history of vesicular lesions in at least 50% of the recurrent episodes of cold sores.
* General good health, without other serious medical conditions and specifically with normal renal and hepatic function, as determined by the patient's account of his/her medical history
* Women of child bearing potential had to use an accepted method of birth control (surgical sterilization; intra-uterine contraceptive device; oral contraceptives; hormone delivery systems such as Norplant® or Depo-Provera injections; a diaphragm in combination with contraceptive cream, jelly, or foam; or a condom in combination with contraceptive cream, jelly or foam). Patients unable or unwilling to use one of the methods of birth control listed above for the duration of the study could not enter the study.
* For women of child-bearing potential, a negative pregnancy test (urine) at screening was required
* Signature on the informed consent document

Exclusion Criteria:

* Previous herpes vaccination
* Patients using topical immunosuppressive agents (including steroids, tacrolimus and pimecrolimus) on or near the face or systemic immunosuppressive agents (including steroids, tacrolimus and pimecrolimus) within 30 days of screening
* Patients known to be immunosuppressed due to underlying disease (e.g. HIV infection) or concomitant treatment (e.g. cancer chemotherapy)
* Recent history of alcohol or drug abuse, which in the opinion of the investigator, could interfere with that study patient's compliance with study requirements
* Significant skin disease such as atopic dermatitis or eczema that would interfere with the assessment of lesions
* Allergy or hypersensitivity to formulations containing acyclovir, penciclovir, famciclovir, and/or other nucleoside analogues
* Women who were lactating or breast feeding
* Had already been randomized once into the study
* Patients who had received an investigational drug in the past four weeks

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Dates: Start 2003-10; Study Completion 2007-07 (Actual)

PRIMARY OUTCOMES:
Time to healing of the primary lesion complex (loss of crust from vesicular [classical] lesions)

SECONDARY OUTCOMES:
safety and tolerability assessed by adverse events (AEs)
resolution of pain / discomfort after short-course regimens
proportion of patients with aborted lesions
time to healing of all vesicular lesions
time to healing of all aborted (non-vesicular) lesions

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals Japan, Study Chair — Novartis Pharmaceuticals